CLINICAL TRIAL: NCT04187963
Title: Effects of Group Physical Therapy on Walking Speed in Patients With Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Ciubean Alina Deniza, Principal investigator, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UniversitateaMFHCluj
Record Dates: First submitted 2019-11-28; First posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: case-control
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group physical therapy (Experimental): Groups of 6 patients and 1 physical therapist for the 1.5 hour physical therapy session
  Interventions: Other: Physical therapy
- Individual physical therapy (Active Comparator): 1.5 hour physical therapy session 1 on 1 (1 patient and 1 physical therapist)
  Interventions: Other: Physical therapy

INTERVENTIONS:
Other: Physical therapy — The rehabilitation protocol for the IPT consisted of cardiovascular warm-up activities, stretching exercises, strengthening exercises, functional, gait and balance training, recreational games and ended with relaxation exercises. In addition, the GPT protocol followed the exact same pattern, except for 5-10 minute breaks for informal socialization between participants, at the beginning of the session, mid-session and at the end of the session.
  Also, both groups had access to external cues, which were applied during a variety of tasks and environmental situations, like gait initiation and termination, heel strike and push-off, sideways and backwards stepping, walking while dual tasking, and walking over various surfaces and long distances.

SUMMARY:
Parkinson disease is a progressive neurologic disorder characterized by motor impairments which alter the walking capacity, and lead to reduced walking speed, decreased stride length and increased double support time. Physical therapy interventions are an important part of the non-pharmacological treatment for Parkinson disease. The purpose of this study was to assess whether there is a different outcome regarding improvement of walking speed, when applying a physical therapy program in an individual or in a group manner.

A prospective, observational, cohort type study on 60 patients with Parkinson disease was carried out between November 2014 - July 2017, in the Clinical Rehabilitation Hospital in Cluj-Napoca, Cluj county, Romania. Patients were randomly divided into 2 groups, and were prescribed either individual (1 patient and 1 physical therapist) or group physical therapy (6 patients and 1 physical therapist). Treatment protocol included 10 sessions of physical therapy, in the same room setting and performed the same routine of exercises, except for the 3 breaks during the sessions in the group therapy for informal socialization. Walking speed was measured by two validated instruments, the 6-minute walk test and the 10-meter walk test, before and after treatment.

Patients with PD could benefit more from a group physical therapy program, as gait speed increased significantly. The group approach facilitates interactions and is cost-effective, as it requires only one therapist and more patients.

DETAILED DESCRIPTION:
The current study was carried out during November 2014 - July 2017, in the Clinical Rehabilitation Hospital in Cluj-Napoca, Cluj county, Romania. A total of 60 subjects diagnosed with typical, idiopathic PD participated in this study.

All patients met the following inclusion criteria: (1) stable medication usage; (2) Hoehn and Yahr stage 2, 3 or 4; (3) ability to walk independently or by using an assistive walking device; (4) age 50 to 70 years; (5) no severe cognitive impairments (Mini-Mental State Examination - MMSE score, ≥24); (6) no other severe neurologic, cardiopulmonary or orthopedic disorders; and (7) not having participated in a PT or rehabilitation program in the previous 2 months.

The patients were randomly divided into 2 treatment groups: group physical therapy -GPT (n=30) and individual physical therapy - IPT (n=30).

Treatment protocol for each group included 10 sessions of physical therapy, each 1.5 hour long, on a daily basis for 2 weeks. All treatment sessions occurred at the same time of day throughout the study, in the morning, 60-90 minutes after intake of pharmaceutical treatment for PD. For the GPT, there were groups of 6 patients, supervised by 1 physical therapist. The group sizes were kept small to promote efficiency and motivation. The patients undertaking IPT were alone with the physical therapist during the sessions. Both groups had their encounters in the same physical therapy room setting.

The rehabilitation protocol for the IPT consisted of cardiovascular warm-up activities, stretching exercises, strengthening exercises, functional, gait and balance training, recreational games and ended with relaxation exercises. In addition, the GPT protocol followed the exact same pattern, except for 5-10 minute breaks for informal socialization between participants, at the beginning of the session, mid-session and at the end of the session.

Also, both groups had access to external cues, which were applied during a variety of tasks and environmental situations, like gait initiation and termination, heel strike and push-off, sideways and backwards stepping, walking while dual tasking, and walking over various surfaces and long distances. There is evidence in the literature to support each of the components contained in the intervention.19-25 In order to facilitate initiation and speed of movement, most activities employed visual and auditory cues as triggers. Visual cues were looking at and follow the therapist's movements in the IPT group or the other group member's movements in the GPT group. A mirror was also used. Auditory cues were music with regular rhythm, and verbal suggestions and reinforcement from the therapist, in the IPT group or the therapist and other participants, in the GPT group.

All patients were evaluated at the beginning and at the end of the physical therapy program. The evaluation included the 6-minute walking test and the 10-meter walking test. Gait speed for each participant was calculated as the ratio between the walked distance and the time unit, and it was measured in meters/seconds.

For each subject, all assessment sessions were performed in the morning, by the same person and all tests were performed in the same order, to control for variations in performance because of medication cycle. All assessments were conducted in the "on" state for the subjects experiencing motor fluctuations.

ELIGIBILITY:
Inclusion Criteria:

* stable medication usage;
* Hoehn and Yahr stage 2, 3 or 4;
* ability to walk independently or by using an assistive walking device;
* age 50 to 70 years;
* no severe cognitive impairments (Mini-Mental State Examination - MMSE score, ≥24);
* no other severe neurologic, cardiopulmonary or orthopedic disorders;
* not having participated in a PT or rehabilitation program in the previous 2 months.

Exclusion Criteria:

* not stable medication usage;
* Hoehn and Yahr stage 1;
* inability to walk independently or by using an assistive walking device;
* age less than 50 and more than 70 years;
* severe cognitive impairments (Mini-Mental State Examination - MMSE score, below 24);
* other severe neurologic, cardiopulmonary or orthopedic disorders;
* having participated in a PT or rehabilitation program in the previous 2 months.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in Walking speed (meters/seconds) | at baseline and after 10 days
  the 6-minute walking test
Change in Walking speed | at baseline and after 10 days
  the 10-meter walking test.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol